CLINICAL TRIAL: NCT06125028
Title: A Pivotal Phase 3 Clinical Trial to Assess the Diagnostic Performance and Safety of [68Ga]Ga-PentixaFor ([68Ga]Ga-PTF), a Positron Emission Tomography (PET) Imaging Agent, Versus [18F]FDG PET/CT Imaging, for Staging of Patients With Confirmed Marginal Zone Lymphoma Exemplary for CXCR4-positive Malignant Lymphomas: a Prospective, International, Multi-center, Comparative, Randomized, Cross-over, Open-label Lymphoma Diagnostic Trial
Brief Title: [68Ga]Ga-PentixaFor-PET Imaging for Staging of Marginal Zone Lymphoma
Acronym: LYMFOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Pentixapharm AG (Industry)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PTF301
Record Dates: First submitted 2023-10-13; First posted 2023-11-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- [68Ga]Ga-PTF PET/CT (Experimental): 150 (+/-50) MBq [68Ga]Ga-PTF will be administered intravenously and PET/CT will be performed
  Interventions: Drug: [68Ga]Ga-PentixaFor
- [18F]FDG PET/CT (Active Comparator): [18F]FDG will be administered once intravenously according to the SMPC and PET/CT will be performed
  Interventions: Drug: [18F]Fluorodeoxyglucose

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — [68Ga]Ga-PTF i.v. injection
  Other Names: [68Ga]Ga-PTF
  Arms: [68Ga]Ga-PTF PET/CT
Drug: [18F]Fluorodeoxyglucose — [18F]FDG i.v. injection.
  Other Names: [18F]FDG
  Arms: [18F]FDG PET/CT

SUMMARY:
This will be a pivotal prospective prospective, international, multi-center, comparative, randomized, cross-over, open-label lymphoma diagnostic trial to assess the diagnostic performance and safety of the positron emission tomography (PET) imaging agent [68Ga]Ga-PTF) , versus [18F]FDG PET/CT imaging, for staging of patients with confirmed marginal zone lymphoma exemplary for CXCR4-positive malignant lymphomas.

ELIGIBILITY:
Inclusion criteria:

All patients must meet all of the following criteria:

1. Signed informed consent from the patient.
2. Patients of either gender, aged ≥ 18 years.
3. Patients with a histologically proven diagnosis of marginal zone lymphoma (MZL) according to the World Health Organization (WHO) classification of lymphoid neoplasms. Patients must have a biopsy-proven nodal, extranodal, or splenic MZL (at the time of enrolment, the CXCR4 expression status will be unknown).
4. Treatment-naïve.
5. Negative pregnancy test in women capable of child-bearing and their agreement to use highly effective contraception for 1 month after the last dose of [68Ga]Ga-PTF and [18F]FDG.
6. For male patients whose partner is of child-bearing potential: The patient is willing to ensure that he and his partner use effective contraception for 1 month after the last dose of [68Ga]Ga-PTF and [18F]FDG.
7. Acceptable organ function, as evidenced by the following laboratory data:

   1. No renal impairment: Estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2or creatinine clearance > 60 mL/min by the Cockcroft-Gault equation or equivalent
   2. Total bilirubin ≤ 1.5 × ULN (upper limit of normal)
   3. Serum albumin ≥ 2.5 g/dL.
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN or ≤ 5 × ULN in the presence of liver metastases
   5. International normalized ratio (INR) < 1.3 or ≤ institutional ULN.
8. Life expectancy ≥ 12 weeks as estimated by the Investigator.
9. The patient must not have undergone any physical or pharmacological intervention with curative or palliative intent between the time of any of the diagnostic measures and the [68Ga]Ga-PTF PET/CT and [18F]FDG PET/CT scan.

Exclusion criteria:

Patients will be excluded if one or more of the following criteria are met:

1. Known hypersensitivity to any active pharmaceutical agent or constituent of the [68Ga]Ga-PTF and/or [18F]FDG investigational products.
2. Inability to lie still for the entire imaging time.
3. Any severe acute or active chronic infection, as judged by the Investigator, at the time of screening or within two months prior to screening that may interfere with the diagnostic properties of [68Ga]Ga-PTF PET/CT and/or [18F]FDG PET/CT imaging.
4. Patients with plasma glucose levels higher than 11 mmol/L or 200 mg/dL prior to [18F]FDG administration.
5. Administration of any anti-cancer therapy within 1 month prior to study entry.
6. Patients with complete resection of all tumor lesion(s).
7. Administration of another investigational medicinal product within 30 days or within 5 terminal elimination half-lives of previous investigational medicinal product, whichever is longer, prior to study entry.
8. Current greater than grade 2 toxicity from any reason, per US-NCI "Common Terminology Criteria for Adverse Events v5.0" (NCI CTCAE 2017) except if tumor-related.
9. Pregnant or breast-feeding women.
10. Concomitant prohibited treatment which may interfere with [68Ga]Ga-PTF PET/CT imaging (systemic corticosteroids) administered within the last 1 month prior to study start.
11. Colony-stimulating factor (CSF) therapy within 5 days prior to [18F]FDG PET/CT examination.
12. Any recent myocardial infarction, stroke, or osteomyelitis within two months prior screening.
13. [18F]FDG PET/CT imaging or [68Ga]Ga-PTF PET imaging performed prior to study entry.
14. Judged by the referring physician as not mentally or as not physically fit to understand and comply with protocol-related interventions and procedures (e.g., medically retarded, body weight > 180 kg for PET scanner).
15. Body weight of less than 48 kg.
16. Any other concurrently active neoplasia, or other disease who could jeopardize study safety or data.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity of [68Ga]Ga-PTF PET/CT imaging vs. [18F]FDG PET/CT imaging in tumor detection | Through study completion, an average of 6 months
Specificity of [68Ga]Ga-PTF PET/CT imaging vs. [18F]FDG PET/CT imaging in tumor detection | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Proportion of patients with additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) compared to pre-PET conventional staging as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with a change in intended patient management due to additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) compared to pre-PET conventional staging as assessed by questionnaires completed by an Independent Committee | Through study completion, an average of 6 months
Inter-observer agreement of local and central assessment in terms of staging | Through study completion, an average of 6 months
Proportion of patients with nodal MZL with additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) compared to pre-PET conventional staging as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with extranodal MZL with additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) compared to pre-PET conventional staging as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with splenic MZL with additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) compared to pre-PET conventional staging as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with nodal MZL with a change in intended patient management due to additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with extranodal MZL with a change in intended patient management due to additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF;[18F]FDG) as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Proportion of patients with splenic MZL with a change in intended patient management due to additional or less lesions detected by each PET/CT imaging agent ([68Ga]Ga-PTF and [18F]FDG) as assessed by questionnaires completed by the referring physicians | Through study completion, an average of 6 months
Diagnostic performance, consisting of sensitivity and specificity, of each PET/CT imaging agent in tumor detection on a region-basis (eyes, ears, nose, throat, liver, spleen, gastrointestinal tract, bone marrow) confirmed by SoT or surrogate SoT | Through study completion, an average of 6 months
Sensitivity of each PET/CT imaging agent in tumor detection on a patient-basis confirmed by SoT or surrogate SoT | Through study completion, an average of 6 months
Positive and negative predictive values (PPV, NPV) of each PET/CT imaging agent to detect tumor on a patient-basis and lesion-basis | Through study completion, an average of 6 months
Detection rate of each PET/CT imaging agent to detect tumor on a patient-basis and lesion-basis confirmed by SoT or surrogate SoT | Through study completion, an average of 6 months
Proportion of patients with additional or less tumoral lesions detected by [68Ga]Ga-PTF PET/CT imaging compared to [18F]FDG PET/CT imaging | Through study completion, an average of 6 months
Inter-reader and intra-reader agreement for tumor detection of each PET/CT imaging agent on a lesion-basis and patient-basis | Through study completion, an average of 6 months
Reproducibility of [68Ga]Ga-PTF PET/CT imaging (reproducibility group) | Through study completion, an average of 6 months
Maximum standardized uptake value (SUVmax), SUVpeak and SUV mean of each PET/CT imaging agent | Through study completion, an average of 6 months
Target-to-background ratio (TBR) of each PET/CT imaging agent | Through study completion, an average of 6 months
Contrast-to-noise ratio (CNR) of each PET/CT imaging agent | Through study completion, an average of 6 months
Signal-to-noise ratio (CNR) of each PET/CT imaging agent | Through study completion, an average of 6 months
Frequency and Severity of Adverse Events for each PET/CT imaging agent | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
Frequency and kind of adverse effects present at the injection site | 2-3 hours after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of the injection site status (which kind of adverse effects have appeared) after the injection of each PET/CT imaging compound
Clinical significance of abnormal results during physical examination | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of physical examination findings
Blood pressure (systolic and diastolic) | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of blood pressure (systolic and diastolic)
Heart or pulse rate | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of heart or pulse rate
RR interval findings/abnormalities | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of findings/abnormalities in the RR interval
PQ interval findings/abnormalities | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of PQ interval findings/abnormalities
QRS complex findings/abnormalities | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of QRS complex findings/abnormalities
QT interval findings/abnormalities | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of QT interval findings/abnormalities
QTc interval findings/abnormalities | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of QTc interval findings/abnormalities
Weight | Prior injection of each PET/CT imaging agent and after injection of each PET/CT imaging agent
  The safety and tolerability for each PET/CT imaging agent will be evaluated by the assessment of patient weight

OTHER OUTCOMES:
Sensitivity of [68Ga]Ga-PTF PET/CT imaging in detecting CXCR4 overexpressing tissue confirmed by a CXCR4 SoT (CXCR4 IHC) | Through study completion, an average of 6 months
  Sensitivity of [68Ga]Ga-PTF PET/CT imaging in detecting CXCR4 overexpressing tissue will be analyzed on a lesion-basis and will be confirmed by a CXCR4 SoT (CXCR4 IHC)
Specificity of [68Ga]Ga-PTF PET/CT imaging in detecting CXCR4 overexpressing tissue | Through study completion, an average of 6 months
  Specificity of [68Ga]Ga-PTF PET/CT imaging in detecting CXCR4 overexpressing tissue will be analyzed on a lesion-basis and will be confirmed by a CXCR4 SoT (CXCR4 IHC)
Receiver-operating-characteristic (ROC) curve analysis | Through study completion, an average of 6 months
Determination of the area under the curve (AUC) | Through study completion, an average of 6 months
Correlation of [68Ga]Ga-PTF uptake in PET and CXCR4 overexpression by IHC | Through study completion, an average of 6 months
Correlation of the Ki-67 proliferation index with CXCR4 overexpression and with SUVmean on a lesion-basis | Through study completion, an average of 6 months
Correlation of the Ki-67 proliferation index with CXCR4 overexpression and with SUVmax on a lesion-basis | Through study completion, an average of 6 months
Rate of non-tumoral CXCR4-positive and CXCR4-negative lesions found in the [68Ga]Ga-PTF PET/CT imaging | Through study completion, an average of 6 months
Percentage of patients with within-patient discordant lesions in terms of CXCR4 expression | Through study completion, an average of 6 months
Positive predictive value (PPV) of [68Ga]Ga-PTF PET/CT imaging for detection of CXCR4 overexpressing tissue | Through study completion, an average of 6 months
Negative predictive value (NPV) of [68Ga]Ga-PTF PET/CT imaging for detection of CXCR4 overexpressing tissue | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Buck, Prof. Dr., Principal Investigator — University Hospital Würzburg, Department of Nuclear Medicine
Locations (12):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU La Timone, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Cochin, Paris
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Würzburg, Würzburg
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - L'IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l, Meldola
  - Ospedale San Raffaele S.r.l., Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No